CLINICAL TRIAL: NCT05379478
Title: An Evaluation of Immune Responses to SARS-CoV-2 Infection or Vaccination
Brief Title: Immune Responses to COVID-19 Infection or Vaccination
Status: Completed | Type: Observational
Sponsor: Aditxt, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: R2020-1002
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — up to 30ml of frozen plasma, serum, and isolated PBMCs will be retained for up to 5 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Unvaccinated, COVID naive: Volunteers with no history of COVID-19 or vaccination. This is an observational study with no intervention
  Interventions: Diagnostic Test: Laboratory assessment of antibody profiles
- Unvaccinated, Convalesced: Volunteers with a history of COVID-19 infection but no COVID-19 vaccination. This is an observational study with no intervention
  Interventions: Diagnostic Test: Laboratory assessment of antibody profiles
- Vaccinated: Volunteers with a history of COVID-19 vaccination. This is an observational study with no intervention
  Interventions: Diagnostic Test: Laboratory assessment of antibody profiles

INTERVENTIONS:
Diagnostic Test: Laboratory assessment of antibody profiles — Antibody profiles will be determined on submitted plasma samples

SUMMARY:
The overall purpose of this observational cohort study is to characterize COVID-specific immune responses to SARS-CoV-2 exposure or COVID vaccination in a real-world setting. Participants will be asked to provide blood samples (either a normal venous blood draw, a few drops of blood obtained with a small finger-stick device, or both), as well as saliva or nasal swab sample at a series of visits. Subjects will receive results of the testing that is approved for routine clinical use (i.e., their AditxtScore), while residual samples from each visit will be stored for future testing. These efforts will support ongoing AditxtScore test development and enhance the effectiveness of its interpretation - aiding efforts to maximize benefits of clinical laboratory testing in the pandemic response.

DETAILED DESCRIPTION:
1. Background and Overview Aditxt, Inc, in collaboration with researchers at Stanford University, has laboratory-developed tests (LDTs) for simultaneously monitoring anti-SARS-COV2 antibodies (IgG, IgA, and IgM) directed against 3 different SARS-CoV-2 antigens (RBD, S1, and NP) as well as assessing SARS-CoV-2 neutralizing antibody activity.

   These tests are currently being offered routinely to the public as the AditxtScoreTM at Aditxt's CLIA certified, CAP accredited clinical laboratory in Richmond, VA. Aditxt also performs these tests for research and development purposes at a facility in Mountain View, CA. The AditxtScore provides an ideal platform for real- world investigations of immune responses to SARS-CoV-2 exposure as well as to the COVID-19 vaccines.

   The overall purpose of this observational cohort study is to characterize COVID-specific immune responses to SARS-CoV-2 exposure or COVID vaccination in a real-world setting. Participants will be asked to provide blood samples (either a normal venous blood draw, a few drops of blood obtained with a small finger-stick device, or both), as well as saliva or nasal swab sample at a series of visits. Subjects will receive results of the testing that is approved for routine clinical use (i.e., their AditxtScore), while residual samples from each visit will be stored for future testing. These efforts will support ongoing AditxtScore test development and enhance the effectiveness of its interpretation - aiding efforts to maximize benefits of clinical laboratory testing in the pandemic response.
2. Objectives • To characterize immune responses (e.g., magnitude/strength and temporal dynamics of antibody generation, class switching, and antibody persistence) following exposure to the SARS-CoV-2 virus or COVID-19 vaccination.

   • To investigate between group (eg vaccine vs. natural exposure) and within group (i.e., individual variation) differences in immune responses.

   • To determine the relationship between AditxtScore components and neutralizing antibody activity and other potential correlates of protection, and to describe possible clinical correlates of immune response characteristics.

   • To support test development activities such as determining appropriate clinical cutpoints, analyte stability, and comparability of results from different sample types (e.g., venous blood draw vs fingerstick blood drop, nasal swab vs. saliva collection). These activities will support refinement of existing tests as well as development of future tests (e.g. COVID-19 specific memory B cell, T cell, and NK cell responses).
3. Study Procedures 3a. Subject Recruitment Subject recruitment will consist primarily of word-of-mouth efforts of study personnel (e.g. friend and family networks) and other interested parties in the local community (e.g. a handful of local physicians). No broad advertising campaign is anticipated, though a study announcement flyer describing the study opportunity will be used to support recruitment efforts. Potential subjects will be directed to call Aditxt to schedule a time to come to the laboratory and learn more about the study.

Anyone with a prior history of SARS-CoV-2 exposure, a possible current infection, or a vaccination history is eligible to participate, in addition to negative controls when needed. Efforts will be made to include a representative mix of ages, genders, and ethnicities.

In the special circumstance that a potential subject would like to participate in the study but is unable to come to either Aditxt location (in Richmond, VA or Mountain View, CA) and has access to a qualified phlebotomist, collection materials can be shipped to a qualified phlebotomist in their area for collections. In this case samples would be shipped overnight to Aditxt for processing. The consent forms and patient questionnaire will be emailed to the participant ahead of time and reviewed with the investigator remotely (e.g., via zoom or phone call), signed, and submitted to Aditxt along with the samples.

3b. Administration of Informed Consent and Protection of Privacy Potential study participants will be taken to a private room at Aditxt's facility in either Richmond, VA or Mountain View, CA and the consent form will be explained to them by a member of the study team. Once all questions are answered, if they choose to participate they will sign the consent form. In a situation where the samples are being collected at a different location, the consent and authorization forms will be emailed to the potential subject, printed, and reviewed with a member of the study team remotely (e.g. via zoom or phone call) until all questions have been answered. The consent documents will then be signed and submitted along with the sample.

Study personnel will then assign the participant a subject number and enter the subjects name, subject number, and date of consent on an electronic enrollment log (in an Excel spreadsheet). The enrollment log will be maintained in a secured location on Aditxt's file server with access restricted only to designated study personnel.

The subjects name and date of birth will be used when performing the "routine" testing at each visit (i.e., the PCR virus test and the antibody tests), and standard clinical reports with their names - appropriate for talking to their regular physicians - will be generated and delivered to the subjects. However, only the subject numbers will be used to identify the patient questionnaires and the sample aliquots stored for future testing.

4c. Completion of Patient Questionnaire Once enrolled, subjects will be provided a brief questionnaire to complete to capture information about demographics, any symptoms that may be related to COVID, any comorbid conditions, and current medications they are taking. A followup questionnaire will be provided at each follow-up visit.

4d. Sample Collection

* Health and Safety Precautions Due to the potential risk of viral transmission, the following safety precautions will be adhered to for every study collection (these are the same precautions required by Aditxt for all routine sample collections)

  - Only one subject will be allowed in the collection area at a time.

  - Proper Personal Protective Equipment (PPE) must always be worn by collection personnel when within 6 feet of the patient. This includes a protective gown, gloves, protective mask and face shield.

  - Patients must wear a protective mask in the collection area except when temperature measurement and nasal swab collection are performed.

  - Laboratory collection personnel will clean the collection seat with a disinfectant wipe between patient collections.

  - After collection and the patient has left the collection area, laboratory collection personnel will change gloves and use hand sanitizer at multiple steps in the removal of PPE as outlined in the Procedure section below to ensure no contamination of touched surfaces, including the protective gown, face shield and protective mask.

  - After removal of PPE, laboratory collection personnel will wash hands with soap and water before starting the next patient collection.
  * Face shields will be cleaned with a disinfectant wipe between every patient collection.
  * Protective masks and gowns may be stored for reuse between patient collections if no contamination of the PPE is observed or suspected.
* Phlebotomy Blood samples will be collected identically to those routinely collected for clinical practice, as described in Aditxt's SOP 6037 Anti-SARS-CoV-2 Phlebotomy Procedure.
* Saliva Participants will be asked to rinse their mouth with water 5 minutes prior to collection. They will be provided with a 3mL tube and asked to fill it (by allowing saliva to pool in their mouths and then spitting it into the tube).
* Nasal Swabs Nasal swab samples will be collected identically to those routinely collected for clinical practice, as described in Aditxt's SOP 6036 SARS-CoV-2 Nasal Swab Collection Procedure.
* Finger-stick

Fingerstick capillary blood collection will be performed as follows:

* Wipe the puncture site (the tip of whichever finger the subject prefers) with an alcohol pad and remove the protective cover from the lancet.
* Position the lancet perpendicularly to the underside of the finger and puncture the skin by gently pressing the lancet against the puncture site until it activates.
* Gently apply pressure to the surrounding tissue. Discard the first drop of blood.
* Hold the finger and capillary tube in a downward position. Touch the tip of the capillary to the blood droplet. The tube will fill automatically due to the capillary effect. Collect 3-4 drops of blood (150-250 microL).
* After blood collection, remove the capillary from the tube, dispose of and apply pressure to the puncture site.
* After collection, invert the tube gently several times.
* Apply band-aid to the puncture site.

  4e. Follow-up Visits Subjects will be encourage to return to Aditxt every 1-2 months for additional sample collection for up to 2 years. An updated questionnaire will be completed by the subject at each follow-up visit. Questionnaire and laboratory data will be stored in the study database and identified only by subject number, allowing for additional studies to be performed on the now deidentified data.

  4f. Laboratory Procedures / Reporting The anti-SARS-CoV-2 antibodies and neutralizing antibody activity will be assessed by the AditxtScoreTM flow cytometry method from Aditx Therapeutics. Antigen/virus testing will be performed on the iAMP COVID-19 system from Atila Biosystems. Clinical laboratory reports describing results of this testing will be provided to subjects (exactly as if they had purchased the testing directly).

Additionally, reporting requirements laid out by the US Department of HHS and the Virginia Department of Health will be complied with. Our approach to reporting all routine results is consistent with FDA guidance (Policy for Coronavirus Disease-2019 Tests During the Public Health Emergency (Revised)). Results of future experimental testing performed on stored samples will be de-identified. Individuals will not be notified of future experimental test results.

AditxtScoreTM

o Novel flow cytometry-based method that allows for simultaneous monitoring of IgG, IgA, and IgM antibodies against 3 different COVID antigens, accompanied with a test for corresponding neutralizing antibody activity

iAMP COVID-19 system (Atila Biosystems)

* Isothermal amplification PCR technology detecting sequences from both the "N" gene and the ORF-1ab gene of the SARS-CoV-2 virus
* Approved for use by the FDA under an EUA Aditxt is currently offering this test service routinely).

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate
* 18 years and older

Exclusion Criteria:

* Refusal or inability to provide informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Community members with history of COVID vaccine, COVID exposure, or negative controls
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Laboratory assessment of SARS-CoV-2 antibody profiles | 2 years
  Antibody profiles consist of quantitative determination of IgG, IgM, and IgA levels to the SARs-CoV-2 spike protein (S), receptor binding domain (RBD), and nucleocapsid protein (NP) by flow cytometry. Also, Neutralizing Antibody (NAb) concentrations were determined with a novel ﬂow cytometry based competitive inhibition assay for the measurement of total neutralizing antibodies to different variants of SARS-CoV-2.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Varvel, PhD, Principal Investigator — Aditxt, Inc.
Locations (1):
- Aditxt, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No